CLINICAL TRIAL: NCT04946422
Title: Big Data Research on the Current Situation and Development Trend of Sports Injury Treatment in China
Brief Title: Chinese Sports Injury Treatment Situation and Development Trend of Big Data Research
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2020142
Record Dates: First submitted 2021-06-25; First posted 2021-06-30 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Sports Injury
MeSH Terms: conditions — Athletic Injuries | interventions — Arthroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sports injury-related injuries: Patients who are discharged from the hospital and diagnosed in accordance with sports injury-related injuries, and those whose service item names in the detailed database contain the keyword "arthroscope". Any one of the above will be included in this topic.
  Interventions: Procedure: Arthroscopy

INTERVENTIONS:
Procedure: Arthroscopy — Discharge diagnosis of patients with sports injury-related injuries

SUMMARY:
This project is planned to be based on the medical insurance database collected by the China Health Insurance Research Association (CHIRA). As a national academic research institution, CHIRA collects medical insurance patient data, covering more than 20 provinces across the country. The data of more than 60 municipalities, provincial capitals, and prefecture-level cities are unique and authoritative in my country. Based on the CHIRA database, big data analysis for Chinese sports medicine patients, starting from the names of medical institutions, admission/discharge diagnosis and classification of medical items, etc., to investigate the development trend of arthroscopic surgery in China and understand my country's arthroscopic diseases The distribution characteristics and changing trends of the quantity.

DETAILED DESCRIPTION:
Sports medicine is a multidisciplinary comprehensive discipline, and is positioned as a secondary discipline in the country. It is a clinical application-based discipline that combines medicine and sports to solve sports-related diseases from a medical perspective. The treatment range is centered on the joints. The main treatment method is arthroscopic technology to solve sports-related injuries. Together with postoperative rehabilitation, the goal is to achieve the greatest recovery of motor function. This project is planned to be based on the medical insurance database collected by the China Health Insurance Research Association (CHIRA). As a national academic research institution, CHIRA collects medical insurance patient data, covering more than 20 provinces across the country. The data of more than 60 municipalities, provincial capitals, and prefecture-level cities are unique and authoritative in my country. Based on the CHIRA database, big data analysis for Chinese sports medicine patients, starting from the names of medical institutions, admission/discharge diagnosis and classification of medical items, etc., to investigate the development trend of arthroscopic surgery in China and understand my country's arthroscopic diseases The distribution characteristics and changing trends of the quantity.

ELIGIBILITY:
Inclusion Criteria:

1. Discharge diagnosis of patients with sports injury-related injuries (ICD codes are M12, M13, M15-M19, M20-M25, M65-67, M70, M71, M75, M76, M94 and S33, S40, S43, S46, S51, S53, S63, S8, S73, S93)
2. Patients whose service item name in the detailed database contains the keyword "arthroscope". Any one of the above will be included in this topic.

Exclusion Criteria:

1. After the data is cleaned, it does not meet the requirements of sports injury patients;
2. The data content contains obvious defects and cannot be backfilled.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Sports trauma patients in the Chinese insured population
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2013-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Use of arthroscopy | 2013-2017
  Calculate the use rate of arthroscopy for various types of sports injuries (arthroscope use rate = number of patients with various types of sports injuries who use arthroscopy/total number of visits for this type of injury) , Get a list of the usage rate of arthroscopy for various sports injuries.

CONTACTS AND LOCATIONS:
Overall Officials: jiakuo yu, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No